CLINICAL TRIAL: NCT04712149
Title: Pilot Study - Measurement of Cost, Outcome and Patient Experience of a Digital Weekly Follow up of Lung Cancer Patients
Brief Title: Pilot Digital Follow-up of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: AZ Delta (Other)
Responsible Party: Principal Investigator, prof. dr. Wim Marneffe, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FU- Lung cancer - 001
Record Dates: First submitted 2020-12-18; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): In the intervention arm, 15 patients will receive a weekly questionnaire. Alerts will be sent to the multidisciplinary care team, who will undertake follow-up actions. In the control arm, 15 patients will receive the standard care pathway without weekly questionnaire and without automatic alerts to the care team. The standard care pathways and the care team are the same in both groups. In this pilot study, the weekly follow-up will be evaluated by a validation questionnaire, semi-structured interviews with patients and the care team, and workload registration of the care team during a six-month period.
  Interventions: Device: Weekly digital follow up
- Control arm (No Intervention)

INTERVENTIONS:
Device: Weekly digital follow up — weekly digital follow-up by sending a questionnaire to patients and sending alerts based on the questionnaire to the care team
  Arms: intervention arm

SUMMARY:
In the pilot study, 30 patients with metastatic lung cancer (stage IV) will be recruited at the start of their stage IV treatment from February 2019. The study period per patient will last six months, from the start of the stage IV treatment. Patients are eligible if they are diagnosed with stage IV lung cancer, speak sufficient Dutch, and are willing to participate. Patients are randomly assigned to two arms by simple randomization. In the intervention arm, 15 patients will receive a weekly questionnaire. Alerts will be sent to the multidisciplinary care team, who will undertake follow-up actions. In the control arm, 15 patients will receive the standard care pathway without weekly questionnaire and without automatic alerts to the care team. The standard care pathways and the care team are the same in both groups. In this pilot study, the weekly follow-up will be evaluated by a validation questionnaire, semi-structured interviews with patients (n=5) and the care team (n=5), and workload registration of the care team during a six-month period for all included patients in the pilot.

ELIGIBILITY:
Inclusion Criteria:

* stage IV lung cancer,
* speak sufficient Dutch
* willing to participate

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Assess the response rates on the digital weekly questionnaire | up to 26 weeks
  In the weekly digital questionnaire the patient reports adverse events and psychosocial support needs. Based on this questionnaire alerts are generated to the care team
Assess the Response on the validation questionnaire at Baseline and at Week 26 | up to 26 weeks
  In the validation questionnaire the patient evaluates the online system, the relevance and difficulty of the questions
Assess the workload of responding to the alerts on the weekly questionnaire for the care team | up to 26 weeks
  the workload is assessed by daily registration of the workload (in minutes) per patient during the six-month registration period by the care team: 2 MD pulmonologists, oncology nurse, psychologist, palliative support, and dietician
Assess the clinical utility of the alerts for the care team | month 6
  In semi-structured interviews with the multidisciplinary care team, the clinical utility of receiving and responding to alerts is assessed with every care giver: an MD pulmonologist, oncology nurse, psychologist, palliative support, and dietician

SECONDARY OUTCOMES:
Validation questionnaire | Baseline
Validation questionnaire | month 6
Weekly questionnaire based on PRO CTC-AE | up to 26 weeks
  As individuals go through treatment for their cancer they sometimes experience different symptoms and side effects. For each question, please select the one response that best describes your experiences over the past 7 days…
EORTC QLQ-C30 | Baseline
  Questionnaire developed to assess the quality of life of cancer patients The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. No item occurs in more than one scale ( range in score from 0 to 100).
EORTC QLQ-C30 | week 6
  Questionnaire developed to assess the quality of life of cancer patients The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. No item occurs in more than one scale ( range in score from 0 to 100).
EORTC QLQ-C30 | week 12
  Questionnaire developed to assess the quality of life of cancer patients The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. No item occurs in more than one scale ( range in score from 0 to 100).
EORTC QLQ-C30 | week 18
  Questionnaire developed to assess the quality of life of cancer patients The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. No item occurs in more than one scale ( range in score from 0 to 100).
EORTC QLQ-C30 | week 24
  Questionnaire developed to assess the quality of life of cancer patients The EORTC QLQ-C30 comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. No item occurs in more than one scale ( range in score from 0 to 100).
QLQ-LC13 | baseline
  The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30). Scale 1-4 (1 Not at all - 4 very much).
QLQ-LC13 | week 6
  The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30). Scale 1-4 (1 Not at all - 4 very much).
QLQ-LC13 | week 12
  The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30). Scale 1-4 (1 Not at all - 4 very much).
QLQ-LC13 | week 18
  The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30). Scale 1-4 (1 Not at all - 4 very much).
QLQ-LC13 | week 24
  The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30). Scale 1-4 (1 Not at all - 4 very much).

CONTACTS AND LOCATIONS:
Overall Officials: Wim Marneffe, prof. dr., Principal Investigator — Hasselt University; Veerle Ross, dr., Study Chair — Hasselt University
Locations (1):
- AZ Delta, Roeselare, Belgium

REFERENCES:
- [Derived] Misplon S, Marneffe W, Himpe U, Hellings J, Demedts I. Evaluation of the implementation of Value-Based Healthcare with a weekly digital follow-up of lung cancer patients in clinical practice. Eur J Cancer Care (Engl). 2022 Nov;31(6):e13653. doi: 10.1111/ecc.13653. Epub 2022 Jul 12. PMID 35819130